CLINICAL TRIAL: NCT02641327
Title: Protocol for Evaluation of EarlySense: A Contact-less Device for Monitoring Changes in Blood Pressure
Brief Title: Monitoring Changes in Blood Pressure
Status: Completed | Type: Observational
Sponsor: EarlySense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ES-CLC-2015_Prot_1_BP
Record Dates: First submitted 2015-12-14; First posted 2015-12-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-09

CONDITIONS: Blood Pressure
Keywords: Inhospital patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Internal ward: Patients hospitalized in Internal Medicine unit with unstable blood pressure that need regulation/ stabilization of their blood pressure (e.g., CHF, post surgical, hypotension or Hypertension patients, patients with kidney failure, heart disease, stroke)
  Interventions: Device: EarlySense (Passive monitoring)
- ICU: Patients hospitalized in intensive care with arterial line that allow continuous blood pressure measurement
  Interventions: Device: EarlySense (Passive monitoring)

INTERVENTIONS:
Device: EarlySense (Passive monitoring) — Passive contact-free monitoring

SUMMARY:
The study objective is to assess the accuracy of Earlysense contactless monitoring to detect changes in blood pressure vs. Gold reference method / devices including ambulatory blood pressure monitoring device (ABPM) or invasive blood pressure monitoring for patients who have arterial line as part of their standard clinical care.

DETAILED DESCRIPTION:
The study objective is to collect data to assess the accuracy and reliability of Earlysense contactless monitoring for blood pressure monitoring vs. gold reference methods such as ABPM (Ambulatory blood pressure measurement) for patients hospitalized in Internal Medicine department and vs. Arterial Line measurements for patients hospitalized in ICU. In addition the collected data will be used to further enhance and improve the existing algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and up
2. Patients hospitalized that require stabilization of his/ her blood Pressure
3. Is willing to sign the consent form.

Group II: Patients hospitalized in Intensive Care

1. Age 18 years and up in intensive care with arterial line that allows invasive Blood Pressure measurements
2. Patient or next of kin or legal guardian are willing to sign consent form

Exclusion Criteria:

1. Age < 18 years
2. Does not sleep on a mattress that allows placing EarlySense sensor under it
3. Patient or next of kin or legal guardian is not willing to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 2 groups will be recruited:
  1. Patients hospitalized in Internal Medicine unit with unstable blood pressure that need regulation/ stabilization of their blood pressure (e.g., CHF, post surgical, hypotension or Hypertension patients, patients with kidney failure, heart disease, stroke)
  2. Patients hospitalized in intensive care with arterial line that allow continuous blood pressure measurement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluate accuracy: Blood pressure measured by the EarlySense system in comparison with Gold Standard Devices | 3 months
  Determine the accuracy of the EarlySense system to measure blood pressure in a contactless way: we would like to see what were the BP measurements in the Gold Standard Devices, compares to what the EarlySense System was measuring at the same time

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Hospital, Holon, Israel

IPD SHARING:
Plan to Share IPD: Undecided